CLINICAL TRIAL: NCT05005572
Title: Treatment Choice and Outcomes for End Stage Renal Disease: Evidence From the First Year of a Nationwide Randomized Evaluation
Brief Title: Treatment Choice and Outcomes for ESRD: Evidence From the First Year of a Nationwide Randomized Evaluation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amy Finkelstein (Other)
Collaborators: Massachusetts Institute of Technology (Other)
Responsible Party: Sponsor-Investigator, Amy Finkelstein, Scientific Director, Abdul Latif Jameel Poverty Action Lab
Organization: Abdul Latif Jameel Poverty Action Lab (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: JPAL-9512
Record Dates: First submitted 2021-08-06; First posted 2021-08-13 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-10

CONDITIONS: End Stage Renal Disease
Keywords: Hemodialysis; Peritoneal Dialysis
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Transplantation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental)
  Interventions: Other: Payment adjustment for home dialysis and transplant
- Control (No Intervention)

INTERVENTIONS:
Other: Payment adjustment for home dialysis and transplant — The ETC model makes two types of payment adjustments for facilities and managing clinicians, an adjustment to the reimbursement rate for home dialysis, and a performance adjustment. The first adjustment, Home Dialysis Payment Adjustment (HDPA), raises the reimbursement rate for home dialysis for the first three years of the program; the amount of increase is 3% in 2021, and reduces to 2% in 2022, and 1% in 2023. The second adjustment, Performance Payment Adjustment (PPA), is an increase or decrease in the reimbursement rate based on the home dialysis rate and the transplant rate attributable to the participating facility or clinician.
  Arms: Treatment

SUMMARY:
The investigators plan to analyze the first year of a nationwide randomized-controlled trial of end stage renal disease (ESRD) treatment choice model (ETC). This mandatory-participation program was designed by the Centers for Medicare and Medicaid Services and randomization was conducted at the hospital referral region (HRR) level. 95 HRRs were assigned to the treatment group beginning in January 2021. The investigators will study the impact of this program in the first year on treatment modality choice for ESRD and explore heterogeneity in impact across patients and providers.

ELIGIBILITY:
Inclusion Criteria:

* All Medicare-certified ESRD facilities and Medicare-enrolled managing clinicians located in HRRs in the United States are required to participate.
* Patient is receiving dialysis or other services for ESRD
* Patient is new to dialysis, defined as not having received dialysis for at least 12 months prior to their first observed dialysis claim
* Patient is enrolled in Medicare Part B

Exclusion Criteria:

* HRRs in US territories
* HRRs with 20% or more zip codes in Maryland (excluded from randomization)
* Facilities and clinicians with fewer than 11 attributed beneficiaries
* Patient is receiving dialysis only for an acute kidney injury
* Patient is younger than 66 years of age before initiating dialysis
* Patient received a kidney transplant within 12 months prior to the start of dialysis and does not have a kidney transplant failure code
* Patient is enrolled in Medicare Advantage, a cost plan, or other Medicare managed care plan
* Patient resides outside of the US or in one of the US territories
* Patient has elected hospice
* Patient has a diagnosis of dementia at any point in the first 90 days or the preceding 12 months before initiating dialysis as identified using Centers for Medicare and Medicaid Services Hierarchical condition categories (CMS-HCC)
* Patient is residing in or receiving dialysis in a skilled nursing facility (SNF)

Min Age: 66 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 18621 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Percentage of Patients Receiving Any Home Dialysis in the First 90 Days | The 90-day period beginning on the date of the first dialysis claim.
  It is defined as the percentage of patients in our baseline sample who have any home dialysis claims within the first 90 days since the start of dialysis treatment.

SECONDARY OUTCOMES:
Percentage of Weeks Receiving Any Home Dialysis in First 90 Days | The 90-day period beginning on the date of the first dialysis claim.
  For each patient, this is the number of weeks the patient received dialysis at home or receiving training for home dialysis within the first 90 days divided by the number of weeks the patient received dialysis in any modality in the first 90 days. For the 13th week since the start of dialysis, only the 6 days that fall within the 90-day period are counted and the week is weighted at 6/7 of the other weeks when computing this measure.
Percentage of Dialysis Sessions at Home in First 90 Days | The 90-day period beginning on the date of the first dialysis claim.
  For each patient, this is the number of dialysis sessions at home divided by the total number of dialysis sessions in the first 90 days, weighting peritoneal dialysis sessions as 3/7 of hemodialysis sessions.

OTHER OUTCOMES:
Dialysis Rate per Capita | 9 months
  This is the number of Traditional Medicare patients aged 66 and above who start dialysis in either modality in our baseline sample divided by the number of Traditional Medicare patients aged 66 and above. Patients are counted at the time they start dialysis.
Total Number of Dialysis Patients | 9 months
  This is the number of Medicare patients who are on dialysis in either modality. All dialysis patients are included when computing this measure, not just new patients.
Pre-Dialysis Elixhauser Index | 1 year before first dialysis session
  This is the average pre-dialysis Elixhauser index among patients in our baseline sample.
Percentage of Patients Receiving Any Home Dialysis in First 90 Days in 2020 | The 90-day period beginning on the date of the first dialysis claim.
  This is defined the same way as our primary outcome, except that outcomes are measured using data from the year prior to ETC (2020).

CONTACTS AND LOCATIONS:
Overall Officials: Amy Finkelstein, PhD, Principal Investigator — Massachusetts Institute of Technology; Liran Einav, PhD, Principal Investigator — Stanford University; Neale Mahoney, PhD, Principal Investigator — Stanford University; Yunan Ji, BA, Principal Investigator — Harvard University
Locations (1):
- Massachusetts Institute of Technology, Cambridge, Massachusetts, United States

REFERENCES:
- [Result] Ji Y, Einav L, Mahoney N, Finkelstein A. Financial Incentives to Facilities and Clinicians Treating Patients With End-stage Kidney Disease and Use of Home Dialysis: A Randomized Clinical Trial. JAMA Health Forum. 2022 Oct 7;3(10):e223503. doi: 10.1001/jamahealthforum.2022.3503. PMID 36206005